CLINICAL TRIAL: NCT07351435
Title: The Caribbean Registry of Extracorporeal Membrane Oxygenation (ECMO) From the University Hospital in Martinique
Status: Not yet recruiting | Type: Observational
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Marc Licker, Honorary Professor at the University of Geneva, Consultant in the department of Cardiothoracic Anesthesia and Critical Care at the University Hospital of Martinique, University of Genova
Other Study IDs: 18-11-2025 CHUM CVT
Record Dates: First submitted 2025-11-18; First posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2025-01

CONDITIONS: Cardiogenic Shock; Malignant Arrhythmias; Ischemic or Valvular Heart Failure; Drepanocytosis and Thoracic Syndrome; Pulmonary Thromboembolisms; Sepsis; ARDS (Acute Respiratory Distress Syndrome); Intoxication; Cardiac Arrest (CA); Postcardiotomy Heart Failure; Acute Respiratory Failure
Keywords: acute heart failure; respiratory insufficiency
MeSH Terms: conditions — Shock, Cardiogenic; Ischemia; Sickle Cell Trait; Pulmonary Embolism; Sepsis; Acute Lung Injury; Heart Arrest; Respiratory Insufficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- VV-ECMO: Patients with respiratory failure
- VA-ECMO: Patients with cardiac failure or combined cardiopulmonary failure
- VAV-ECMO: Patients initially on VV or VA-ECMO who require additional respiratory/circulatory support

SUMMARY:
The project's main goal is to collect baseline clinical and procedural data as well as to assess clinical outcomes for all patients undergoing VV, VA or VAV ECMO implantation in the French West Indies and Guiana. All patients undergoing ECMO implantation will be prospectively registered.

DETAILED DESCRIPTION:
In the Caribbean region, access to advanced cardiac interventions faces difficulties owing to unequal distribution of health care resources, medical shortages and distance between health care centers in various islands.

At the University Hospital of Martinique (UHM) in Fort de France, a mobile ECMO team is available 24h a day, 7 days a week, for cardiopulmonary mechanical support in the French Overseas Territories and neighboring islands.

Implantation of veno-venous or veno-arterial (VV or VA) ECMO can be performed at the UHM or at remote hospitals. Some patients on VA-ECMO are transfered by airflight to the UHM and/or to French mainland whenever cardiac transplantation is indicated.

Since 2010, the ECMO-UHM database is a prospective event-driven registry housed and updated by the HeartTeam (perfusionnists, emergency and ICU physicians, cardiac surgeons, cardiothoracic anesthesiologists, cardiologists).

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients implanted with a veno-venous extracorporeal membrane oxygenation device or extracorporeal membrane oxygenation device by the HeartTeam from the University Hospital of Martinique (UHM) from January 2010

Exclusion Criteria:

* Patients with incomplete data (primary endpoint and less than 80% secondary study outcomes)

Max Age: 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients implanted with a VV-ECMO, VA-ECMO or VAV-ECMO device by the UHM HeartTeam
Sampling Method: Non-Probability Sample
Enrollment: 1200 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2032-12-31 (Estimated); Study Completion 2033-06-30 (Estimated)

PRIMARY OUTCOMES:
Mortality at 30 days | from canula implantation to 30 days afterwards
  Number of deceased participants as assessed at 30 days after ECMO implantation

SECONDARY OUTCOMES:
Number of participants with major adverse events | From canula implantation to up to 6 months after ECMO implantation
  Major Adverse events (AE; numbers and rates) as assessed by the consensus statement of the mechanical circulatory support academic research consortium

CONTACTS AND LOCATIONS:
Overall Officials: Marc LICKER, BC, Principal Investigator — CHU Martinique

IPD SHARING:
Plan to Share IPD: Yes
only IPD used in the results publication
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: from January 2026 to December 2032

REFERENCES:
- [Background] Serpa Neto A, Higgins AM, Bailey MJ, Anderson S, Bernard S, Fulcher BJ, Jones A, Linke NJ, Board JV, Brodie D, Buhr H, Burrell AJC, Cooper DJ, Fan E, Fraser JF, Gattas DJ, Hopper IK, Huckson S, Litton E, McGuinness SP, Nair P, Orford N, Parke RL, Pellegrino VA, Pilcher DV, Dicker C, Reddi BAJ, Stub D, Trapani TV, Udy AA, Hodgson CL; EXCEL Study Investigators on behalf of the International ECMO Network (ECMONet). Long-Term Functional Outcomes in the First 12 Months After VA-ECMO in Adult Patients: A Prospective, Multicenter Study. Circ Heart Fail. 2025 Jun;18(6):e012476. doi: 10.1161/CIRCHEARTFAILURE.124.012476. Epub 2025 Apr 29. PMID 40298907
- [Background] Ling RR, Chen Y, Low CJW, Agerstrand C, Jung JS, Lim SL, Lorusso R, Mueller T, Okada Y, Tonna JE, Shekar K, Brodie D, MacLaren G, Ramanathan K. Left ventricular unloading during extracorporeal cardiopulmonary resuscitation: a target trial emulation of the ELSO registry. Crit Care. 2025 May 8;29(1):186. doi: 10.1186/s13054-025-05345-3. PMID 40340843
- [Background] Grazioli A, Plazak M, Willsey K, Rabin J, Rector RP, Belyayev L, Lankford AS, Scalea TM, Shah A, Taylor BS, Gladwin MT. Outcomes and survival prediction in adults with sickle cell disease treated with extracorporeal membrane oxygenation. Blood Adv. 2025 Oct 14;9(19):4881-4890. doi: 10.1182/bloodadvances.2025016368. PMID 40644625
- [Background] Labrada L, Alarfaj M, Tran L, Granger H, Hernandez A, Hu J, Baker J, Grandin EW, Delgado AA, Katz JN, Miller PE, Alviar CL, Osborn E, Bacchetta MD, Lindenfeld J, Shah Z, Rali AS. Optimal ECLS Support in Mixed Cardiogenic and Septic Shock: An ELSO Registry Analysis. JACC Adv. 2025 Oct;4(10 Pt 1):101965. doi: 10.1016/j.jacadv.2025.101965. Epub 2025 Jul 23. PMID 40704940
- [Background] Wang L, Wang K, Wang Y, Yang F, Li C, Hao X, Du Z, Rycus PT, Tonna JE, Fan E, Wang H, Hou X. A simple VA-ECMO bundle in adult patients with cardiogenic shock: an analysis of ELSO registry. EClinicalMedicine. 2025 Aug 7;87:103423. doi: 10.1016/j.eclinm.2025.103423. eCollection 2025 Sep. PMID 40823501
- [Background] Baldetti L, Pontillo D, Capoccia M, Kowalewski M, Tonna JE, Broman M, Conrad SA, Swol J, Scandroglio AM, Brewer JM, Maybauer MO, Lorusso R. Venopulmonary extracorporeal life support: An Extracorporeal Life Support Organization registry analysis. J Heart Lung Transplant. 2026 Jan 6:S1053-2498(25)02480-5. doi: 10.1016/j.healun.2025.12.024. Online ahead of print. PMID 41506589
- [Background] Moynihan KM, Sharma M, Mehta A, Lillie J, Ziegenfuss M, Festa M, Chan T, Thiagarajan R. Race-Conscious Research Using Extracorporeal Life Support Organization Registry Data: A Narrative Review. ASAIO J. 2024 Sep 1;70(9):721-733. doi: 10.1097/MAT.0000000000002206. Epub 2024 Apr 18. PMID 38648078
- [Background] Remy T, Jegard J, Chenouard A, Maminirina P, Liet JM, Couec ML, Joram N, Bourgoin P. Characteristics and outcomes of children and young adults with sickle cell disease supported with extracorporeal membrane oxygenation (ECMO): An updated analysis of the ELSO registry. Artif Organs. 2025 Mar;49(3):508-515. doi: 10.1111/aor.14880. Epub 2024 Oct 3. PMID 39360897
- [Background] Mazzeffi M, Zaaqoq A, Curley J, Buchner J, Wu I, Beller J, Teman N, Glance L. Survival After Extracorporeal Cardiopulmonary Resuscitation Based on In-Hospital Cardiac Arrest and Cannulation Location: An Analysis of the Extracorporeal Life Support Organization Registry. Crit Care Med. 2024 Dec 1;52(12):1906-1917. doi: 10.1097/CCM.0000000000006439. Epub 2024 Oct 9. PMID 39382377
- [Background] Kanwar MK, Shah P, Cascino T, Grinstein J, Goldstein D, Hernandez-Montfort J, Li S, Uriel N, Molina E, Cantor R, Komanduri B, Pagani FD, Kirklin JK. Impact of Preoperative Temporary Mechanical Circulatory Support on Durable LVAD Outcomes: An Analysis of The Society of Thoracic Surgeons National Intermacs Database. JACC Heart Fail. 2025 Nov;13(11):102671. doi: 10.1016/j.jchf.2025.102671. Epub 2025 Oct 8. PMID 41193107